CLINICAL TRIAL: NCT05391308
Title: Overnight Rostral Fluid Shift in the Pathogenesis of Obstructive Sleep Apnea in Spinal Cord Injured Patients
Brief Title: Overnight Upper Airway Infiltration in Spinal Cord Injury
Acronym: OUI-SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220159; 2022-A00105-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea; Spinal Cord Injuries
Keywords: Obstructive Sleep Apnea; spinal cord injury; Neck circumference; Neck volume; Fluid shift; Pathophysiology
MeSH Terms: conditions — Sleep Apnea, Obstructive; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): All patients will have pre-polysomnographie and post-polysomnographie mesurement.
  Interventions: Other: Pre-polysomnography mesurement; Other: Polysomnography measure; Other: Post-polysomnography measurements

INTERVENTIONS:
Other: Pre-polysomnography mesurement — Leg fluid volume (bioelectrical impedance), neck circumference (tape measure), neck volume (3D scanner), time spent sitting down (self-reporting)
Other: Polysomnography measure — Apnea-Hypopnea Index
Other: Post-polysomnography measurements — Leg fluid volume (bioelectrical impedance), neck circumference (tape measure), neck volume (3D scanner)

SUMMARY:
Obstructive Sleep Apnea (OSA), a common disorder resulting from repetitive pharyngeal collapse during sleep, is multifactorial. Usually, OSA is considered primarily a problem of upper airway anatomy, with the craniofacial structure or neck fat decreasing the size of the pharyngeal airway lumen. Obesity, male sex and genetics are well established pathogenic factors. In the last decade rostral fluid displacement (fluid shift) to explain the pathogenesis of upper airway collapsibility has been increasingly studied.

Individuals living with spinal cord injury are at increased risk for OSA, with a prevalence that is three- to fourfold higher than the general population. Individual with acute tetraplegia and undiagnosed or untreated OSA may participate less in rehabilitation due to sleepiness and fatigue and therefore be less engaged in activities that improve quality of life and maintain functioning over time. Intermittent hypoxia, sleep fragmentation and alterations of the autonomous nervous system induced by OSA are thought to delay or limit recovery and in the long term, increase cardio- and cerebrovascular morbi-mortality.

Redolfi et al have shown that overnight change in leg fluid volume correlated strongly with the Apnea Hypopnea index (AHI) and the time spent sitting. In SCI patients two mechanisms may underline fluid shift importance in the pathogenesis of OSA: first, time spent sitting is obviously increased in patients with no walking abilities (prolonged sitting position in wheelchair). Secondly, motor deficit lead to the loss of skeletal muscle pumping activity which could promote leg fluid accumulation during the day.

In our knowledge, no study has specifically assessed the impact of rostral fluid displacement on upper airway collapsibility among patients with spinal cord injury.

Better comprehension of upper airway collapsibility determinants in patients with spinal cord injury is mandatory to identify new therapeutic targets (diuretics, contention…) especially since CPAP, the first line treatment for severe OSA, continue to pose adherence issues in SCI patients. In the future, phenotyping OSA patients, especially those with SCI, will improve personalized management.

The main objective is to find if there is a correlation between the apnea-hypopnea index (AHI) and rostral fluid shift overnight, in non-obese spinal cord injured patients. The secondary aim is to find if there is a correlation between AHI and:

* Neck circumference
* Neck volume
* Time spent sitting down

DETAILED DESCRIPTION:
All SCI patients meeting inclusion criteria with scheduled polysomnography within the framework of usual care and referred to the sleep laboratory will be proposed to participate. These patients are usually recorded in a dedicated room within PMR units during a 3-day to one-week hospital stay.

Information will be given to eligible patients to allow time for reflexion before written consent is collected during the inclusion visit (during the PMR hospitalization or at the sleep laboratory to carry out the night recording).

Collection of clinical and demographic data will be performed by a PMR practitioner or sleep physician according to a predefined and standardized evaluation grid.

After consent form signature patients willing to participate will undergo "before-sleep" measurement of:

* Leg fluid volume
* Neck circumference
* Neck volume
* Short questionnaire developed for the needs of the study. Then patients will undergo a full night polysomnography according to the American Academy of sleep Medicine (AASM) guidelines.

The sleep recording will be carried out in a dedicated room within the spinal cord injury unit with the immediate proximity of a care team with specific competence in the field of the management of the heaviest patients (e.g: urinary catheterization, stool evacuation, pressure sore prevention, safe transfers, etc.).

The reading of the polysomnography will be ensured by a doctor specialized in sleep pathologies without any knowledge of the different impedance measurements, circumference and cervical volume measurements.

"After-sleep" measurement will be performed immediately after patients awakening (before any wheelchair transfer):

* Leg fluid volume
* Neck circumference
* Neck volume
* Short questionnaire developed for the needs of the study.

In summary: Before going to bed and before getting up for the first time, each patient will benefit from a standardized evaluation by measuring bioelectrical impedance on the lower limbs, 3D cervical acquisition and measurement of the neck circumference.

All of these measurements are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

Specific criteria:

* Low cervical (< C6), thoracic or lumbar traumatic spinal cord injury (SCI);
* BMI < 30Kg/m² ;
* Clinically complete SCI (AIS A) or incomplete with no walking ability;
* Neurological level;
* Aged >18 years;
* Patients with a previous indication for polysomnography as part of routine care and referred to sleep laboratory.

No-specific criteria:

* Affiliated to the social security system;
* Absence of serious intercurrent event.

Exclusion Criteria:

Specific criteria:

* Lower limbs amputation ;
* Treated OSA;
* Ongoing diuretic treatment;
* Pregnant woman;
* Pacemaker or other (spinal) stimulation equipment.

No-specific criteria:

* Patient refusal;
* Patient in a period of exclusion from another protocol;
* Inability to sign informed consent;
* Medical or surgical emergency context;
* Vulnerable person or adult subject to legal protection: pregnant or lactating women, person deprived of their liberty by judicial or administrative decision, person hospitalized without consent, or admitted for purposes other than research, Articles L1121 -5 to L1121-8.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between Apnea-Hypopnea Index (polysomnography) and the overnight change in leg fluid volume (bioelectrical impedance) | 18 hours
  AHI is used to diagnose OSA by counting respiratory events. An index greater than 5 per hour defines a ventilatory disorder.
  AHI defines severity as well, the index is:
  * Mild, between 5 and 15 per hour
  * Moderate, between 15 and 30 per hour
  * Severe, over than 30 per hour Leg fluid volume is measured by bioelectrical impedance before and after the night of polysomnography. Intra- and extracellular water are measured in L. Patient is lying down during the measure.

SECONDARY OUTCOMES:
Correlation coefficient between Apnea-Hypopnea Index (polysomnography) and change in neck circumference (tape measure) | 18 hours
  AHI is used to diagnose OSA by counting respiratory events. An index greater than 5 per hour defines a ventilatory disorder.
  AHI defines severity as well, the index is:
  * Mild, between 5 and 15 per hour
  * Moderate, between 15 and 30 per hour
  * Severe, over than 30 per hour Neck circumference is measured by tape measure before and after the night of polysomnography. The circumference is measured at the superior border of the cricothyroid cartilage. The measure is in cm. Patient is lying down during the measure.

OTHER OUTCOMES:
Tertiary outcome: Correlation coefficient between Apnea-Hypopnea Index (polysomnography) and change in neck volume (3D scanner) | 18 hours
  AHI is used to diagnose OSA by counting respiratory events. An index greater than 5 per hour defines a ventilatory disorder.
  AHI defines severity as well, the index is:
  * Mild, between 5 and 15 per hour
  * Moderate, between 15 and 30 per hour
  * Severe, over than 30 per hour Neck volume is recovered through the analysis of images made with the 3D scanner, before and after the night of polysomnography. Volume is in mm3. Patient is lying down during the measure.
Quaternary outcome: Correlation coefficient between Apnea-Hypopnea Index (polysomnography) and time spent sitting down | 18 hours
  AHI is used to diagnose OSA by counting respiratory events. An index greater than 5 per hour defines a ventilatory disorder.
  AHI defines severity as well, the index is:
  * Mild, between 5 and 15 per hour
  * Moderate, between 15 and 30 per hour
  * Severe, over than 30 per hour Time spent sitting down the day of polysomnography is self-reported by patient. Sitting time is in hour and minute.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LEOTARD, MD, Principal Investigator — Unité des pathologies du sommeil, Service de physiologie explorations fonctionelles, Hôpital Raymond Poincaré, APHP
Locations (1):
- Unité des pathologies du sommeil, Service de physiologie explorations fonctionelles, Hôpital Raymond Poincaré, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Redolfi S, Yumino D, Ruttanaumpawan P, Yau B, Su MC, Lam J, Bradley TD. Relationship between overnight rostral fluid shift and Obstructive Sleep Apnea in nonobese men. Am J Respir Crit Care Med. 2009 Feb 1;179(3):241-6. doi: 10.1164/rccm.200807-1076OC. Epub 2008 Nov 14. PMID 19011149
- [Background] Sankari A, Vaughan S, Bascom A, Martin JL, Badr MS. Sleep-Disordered Breathing and Spinal Cord Injury: A State-of-the-Art Review. Chest. 2019 Feb;155(2):438-445. doi: 10.1016/j.chest.2018.10.002. Epub 2018 Oct 12. PMID 30321507
- [Background] Panza GS, Sutor T, Gee CM, Graco M, McCully KK, Chiodo A, Badr MS, Nash MS; American Congress of Rehabilitation Medicine, Interdisciplinary Special Interest Group, Spinal Cord Injury Physical Function and Wellness Task Force. Is Sleep Disordered Breathing Confounding Rehabilitation Outcomes in Spinal Cord Injury Research? Arch Phys Med Rehabil. 2022 May;103(5):1034-1045. doi: 10.1016/j.apmr.2021.08.015. Epub 2021 Sep 17. PMID 34537222
- [Background] Bailly S, Grote L, Hedner J, Schiza S, McNicholas WT, Basoglu OK, Lombardi C, Dogas Z, Roisman G, Pataka A, Bonsignore MR, Pepin JL; ESADA Study Group. Clusters of sleep apnoea phenotypes: A large pan-European study from the European Sleep Apnoea Database (ESADA). Respirology. 2021 Apr;26(4):378-387. doi: 10.1111/resp.13969. Epub 2020 Nov 2. PMID 33140467
- [Background] Proserpio P, Lanza A, Sambusida K, Fratticci L, Frigerio P, Sommariva M, Stagni EG, Redaelli T, De Carli F, Nobili L. Sleep apnea and periodic leg movements in the first year after spinal cord injury. Sleep Med. 2015 Jan;16(1):59-66. doi: 10.1016/j.sleep.2014.07.019. Epub 2014 Oct 7. PMID 25454844
- [Background] Popa C, Popa F, Grigorean VT, Onose G, Sandu AM, Popescu M, Burnei G, Strambu V, Sinescu C. Vascular dysfunctions following spinal cord injury. J Med Life. 2010 Jul-Sep;3(3):275-85. PMID 20945818
- [Background] Redolfi S, Arnulf I, Pottier M, Lajou J, Koskas I, Bradley TD, Similowski T. Attenuation of obstructive sleep apnea by compression stockings in subjects with venous insufficiency. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1062-6. doi: 10.1164/rccm.201102-0350OC. PMID 21836140
- [Background] Murata J, Murata S, Yamagata S, Ohyama M, Kogo H, Umeki N. The attenuating effect of a dynamic cushion on the development of leg edema in wheelchair users with spinal cord injuries. Technol Health Care. 2020;28(4):447-452. doi: 10.3233/THC-192045. PMID 31958103
- [Background] Viaene A, Roggeman S, Goessaert AS, Kessler TM, Mehnert U, Besien VV, De Muynck M, Everaert K. Conservative treatment for leg oedema and the effect on nocturnal polyuria in patients with spinal cord injury. BJU Int. 2019 May;123(5A):E43-E50. doi: 10.1111/bju.14672. Epub 2019 Feb 6. PMID 30653810
- [Background] Leotard A, Levy J, Perennou D, Pepin JL, Lofaso F, Bensmail D, Lebret M, Baillieul S. Sleep might have a pivotal role in rehabilitation medicine: A road map for care improvement and clinical research. Ann Phys Rehabil Med. 2021 Jul;64(4):101392. doi: 10.1016/j.rehab.2020.04.006. Epub 2020 Oct 14. No abstract available. PMID 32445976
- [Background] Berry RB, Brooks R, Gamaldo C, Harding SM, Lloyd RM, Quan SF, Troester MT, Vaughn BV. AASM Scoring Manual Updates for 2017 (Version 2.4). J Clin Sleep Med. 2017 May 15;13(5):665-666. doi: 10.5664/jcsm.6576. No abstract available. PMID 28416048
- [Background] Kaminska M, Jobin V, Mayer P, Amyot R, Perraton-Brillon M, Bellemare F. The Epworth Sleepiness Scale: self-administration versus administration by the physician, and validation of a French version. Can Respir J. 2010 Mar-Apr;17(2):e27-34. doi: 10.1155/2010/438676. PMID 20422065